CLINICAL TRIAL: NCT04808388
Title: Using MRI to Quantify Fatty Infiltration in Muscle Tissue, and Compare it to Isometric Muscle Strength Measurements and (2) Use Questionnaires, Systemic Interview and Simple Myotonic Bed-side Tests to Describe the Phenotype.
Brief Title: Using MRI in Patients With Non-dystrophic Myotonia to Access Muscle Contractility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jonas Jalili Pedersen, Student, Rigshospitalet, Denmark
Other Study IDs: H-18023049(2)
Record Dates: First submitted 2021-03-15; First posted 2021-03-22 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Paramyotonia Congenita; Nondystrophic Myotonia
MeSH Terms: conditions — Myotonic Disorders; Nondystrophic myotonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Using MRI for fat fraction and Biodex for isometric strength

SUMMARY:
The aim of this project is (1) to investigate whether or not structural muscle abnormalities could be a consequence of the disorder and (2) to provide further clinical description of this rare phenotype. To do so, the investigators will (1) use Dixon MRI to quantify fatty infiltration in muscle tissue and compare it to muscle strength measurements from isometric dynamometry in order to access contractility and (2) describe the myotonic phenotype with simple squeeze test and questionnaires.

DETAILED DESCRIPTION:
Non-dystrophic myotonias are rare genetic diseases in which the membrane excitability is altered by mutations in genes encoding muscle ion channels.

Patients suffer from myotonic stiffness, pain, fatigue and sometimes paralysis. Non-dystrophic myotonia is distinct from myotonic dystrophies with the absence of muscle degeneration.

Paramyotonica congenita is characterzied by paradoxial myotonia, which, in contrast to the more common myotonia congenita, is myotonic stiffness that worsens with activity. Typically, the first few contractions seem normal, whereas repetition leads to severe stiffness. Our hypophysis is that these patient might also suffer from muscle degeneration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diagnosed with non-dystrophic myotonia

Exclusion Criteria:

* MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Paramyotonia congenita (prevalence 50-100)
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Contractile properties | 1 year
  Contractility = strength (kg) divided with cross sectional area of the muscle (CCSA)

SECONDARY OUTCOMES:
Muscle strength | 1 year
  Peak torque (maximal contraction in kg) accessed from isometric dynamometry
Cross sectional area (CCSA) | 1 year
  By using MRI to visualize the muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Center Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pedersen JJ, Stemmerik MG, Jacobsen LN, Skriver SV, Wilms GR, Duno M, Vissing J. Muscle fat replacement and contractility in patients with skeletal muscle sodium channel disorders. Sci Rep. 2023 Feb 13;13(1):2538. doi: 10.1038/s41598-023-29759-7. PMID 36782059